CLINICAL TRIAL: NCT02388737
Title: A Randomized, Double-Blind, Double-Dummy, Parallel-group Phase 3 Study to Evaluate the Efficacy and Safety of Oral Once-Daily Administration of TAK-438 10 or 20 mg Compared to Lansoprazole 15 mg in the Maintenance Treatment of Subjects With Endoscopic Healing of Erosive Esophagitis
Brief Title: Efficacy and Safety of Vonoprazan Compared to Lansoprazole in the Maintenance Treatment of Erosive Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-438_305; U1111-1136-5706 (Registry Identifier: WHO); CTR20150039 (Registry Identifier: SFDA CTR)
Record Dates: First submitted 2015-03-09; First posted 2015-03-17 (Estimated); Results first posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Erosive Esophagitis
Keywords: Drug therapy
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vonoprazan 10 mg (Experimental): Lansoprazole 30 mg, capsules or tablets, orally, once, daily, for up to 4 or 8 weeks or until confirmed healing of erosive esophagitis (EE) in healing phase for participants with ongoing EE.
  Vonoprazan 10 mg, tablets, orally, once, daily, and Vonoprazan 20 mg, placebo-matching tablets, orally, once, daily, and Lansoprazole 15 mg placebo-matching, capsules, orally, once, daily, for up to 24 weeks in maintenance phase for participants with confirmed EE healing.
  Interventions: Drug: Vonoprazan; Drug: Lansoprazole; Drug: Vonoprazan Placebo; Drug: Lansoprazole Placebo
- Vonoprazan 20 mg (Experimental): Lansoprazole 30 mg, capsules or tablets, orally, once, daily, for up to 4 or 8 weeks or until confirmed healing of erosive esophagitis (EE) in healing phase for participants with ongoing EE.
  Vonoprazan 20 mg, tablets, orally, once, daily, and Vonoprazan 10 mg, placebo-matching tablets, orally, once, daily, and Lansoprazole 15 mg, placebo-matching capsules, orally, once, daily, for up to 24 weeks in maintenance phase for participants with confirmed EE healing
  Interventions: Drug: Vonoprazan; Drug: Lansoprazole; Drug: Vonoprazan Placebo; Drug: Lansoprazole Placebo
- Lansoprazole 15 mg (Active Comparator): Lansoprazole 30 mg, capsules or tablets, orally, once, daily, for up to 4 or 8 weeks or until confirmed healing of erosive esophagitis (EE) in healing phase for participants with ongoing EE.
  Lansoprazole 15 mg, capsules, orally, once, daily, and Vonoprazan 10 mg, placebo-matching tablets, orally, once, daily, and Vonoprazan 20 mg, placebo-matching tablets, orally, once, daily, for up to 24 weeks in maintenance phase for participants with confirmed EE healing.
  Interventions: Drug: Lansoprazole; Drug: Vonoprazan Placebo

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan tablets
  Other Names: TAK-438
  Arms: Vonoprazan 10 mg; Vonoprazan 20 mg
Drug: Lansoprazole — Lansoprazole capsules or tablets
  Other Names: Prevacid
Drug: Vonoprazan Placebo — Vonoprazan placebo-matching tablets
Drug: Lansoprazole Placebo — Lansoprazole placebo-matching capsules
  Arms: Vonoprazan 10 mg; Vonoprazan 20 mg

SUMMARY:
This is a comparative study of vonoprazan (TAK-438) (10 mg or 20 mg) in participants in whom endoscopic healing of erosive esophagitis has been confirmed with vonoprazan or adequate treatment with a proton pump inhibitor (PPI), to demonstrate the non-inferiority of vonoprazan to lansoprazole in their maintenance treatment (6 months or 24 weeks) as well as to determine the clinically recommended dose for vonoprazan for maintenance therapy in erosive esophagitis.

DETAILED DESCRIPTION:
The drug being tested in this study is called vonoprazan. Vonoprazan is being tested as a maintenance treatment for people with healed erosive esophagitis (EE). This study will look at participants in whom endoscopic healing of erosive esophagitis has been confirmed with vonoprazan or adequate treatment with a proton pump inhibitor (PPI), to demonstrate the non-inferiority of vonoprazan to Lansoprazole in their maintenance treatment (6 months or 24 weeks) as well as to determine the clinically recommended dose for vonoprazan for maintenance therapy in erosive esophagitis.

The study will enroll approximately 693 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the three treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* TAK-438 10 mg
* TAK-438 20 mg
* Lansoprazole 15 mg

Participants with ongoing erosive esophagitis (EE) will receive lansoprazole 30 mg once daily for 4 or 8 weeks (the Healing phase) until healing of EE is confirmed by endoscopy performed at either Week -4 and/or Day 1 before eligible for randomization to maintenance phase. In Maintenance phase, participants with confirming EE healing will be asked to take 2 tablets and a capsule at the same time each morning after breakfast throughout the study. All participants will be asked to record daytime and nighttime (during sleep) subjective symptoms in a diary on a daily basis.

This multi-centre trial will be conducted worldwide. The overall time to participate in this study is 8 months. Participants will make multiple visits to the clinic, and will be contacted by telephone 7-14 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Has been confirmed on endoscopy to have had erosive esophagitis [Los Angeles (LA) classification grades A to D] within 84 days of Day 1.
4. If the participant is not rolled over from TAK-438_303 study, he/she has undergone an open-label Proton pump inhibitor (PPI) treatment (Lansoprazole 30 mg, once daily) of 4 or 8 weeks within the TAK-438_305 protocol.
5. Has been confirmed on endoscopy to have healing of erosive esophagitis. This endoscopy, if not part of the TAK-438_303 study, must have been within the last 14 days prior to randomization, otherwise the endoscopy must be repeated to confirm healing before randomization in the TAK-438_305 study.
6. Is aged 18 years old or older (or the local age of consent if that is older), male or female, at the time of signing an informed consent, and is being treated on an outpatient basis for erosive esophagitis, including those temporarily admitted for examination.
7. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 4 weeks after last dose of study medication.

Exclusion Criteria:

1. Has received any investigational compound (other than study TAK-438_303) within 84 days prior to screening phase.
2. Has received TAK-438 in a previous clinical study (other than study TAK-438_303) or as a therapeutic agent.
3. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Has, in the judgment of the investigator, clinically significant abnormal hematological parameters of hemoglobin, hematocrit, or erythrocytes at Screening.
5. Has a history or clinical manifestations of significant central nervous system (CNS), cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urological, endocrine or hematological disease.
6. Has a history of hypersensitivity or allergies to TAK-438 or to proton pump inhibitors (PPIs) including any associated excipients.
7. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the start the screening phase.
8. Is required to take excluded medications.
9. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
10. Has participated in another clinical study (other than study TAK-438_303) within the past 30 days from Visit 1.
11. Has co-morbidities that could affect the esophagus (eosinophilic esophagitis, esophageal varices, scleroderma, viral or fungal infection, esophageal strictures), a history of radiotherapy or cryotherapy for the esophagus; those with corrosive or physiochemical injury (with the possible inclusion in the study of those with Schatzki's ring or Barrett's esophagus).
12. Has a history of surgical procedures that may affect the esophagus (eg, fundoplication and mechanical dilatation for esophageal strictures excluding Schatzki's ring) or a history of gastric or duodenal surgery excluding endoscopic removal of benign polyps.
13. Developed acute upper gastrointestinal bleeding, gastric ulcer (a mucosal defect with white coating) or duodenal ulcer (a mucosal defect with white coating), within 30 days before the start of the Screening Phase (Visit 1) (with the possible inclusion of those with gastric or duodenal erosion). Participants requiring non-steroidal anti-inflammatory drugs (NSAIDs) or aspirin treatment along with the concomitant PPI therapy to prevent gastrointestinal (GI) bleeding should not be enrolled.
14. Has Zollinger-Ellison syndrome or gastric acid hypersecretion or a history of gastric acid hypersecretion.
15. Is scheduled for surgery that requires hospitalization or requires surgical treatment during his/her participation in the study.
16. Has a history of malignancy or was treated for malignancy within 5 years before the start of the Screening Phase (visit 1) (the participant may be included in the study if he/she has cured cutaneous basal cell carcinoma or cervical carcinoma in situ).
17. Has acquired immunodeficiency syndrome (AIDS) or hepatitis, including hepatitis virus carriers (hepatitis B surface antigen [HBsAg] or hepatitis C virus (HCV)-antibody-positive) (the participant may be included in the study if he/she is HCV-antigen or HCV-ribonucleic acid [RNA]-negative).
18. Laboratory tests performed on visit 1 revealed any of the following abnormalities in the participant:

    1. Creatinine levels: >2 mg/dL (>177 μmol/L).
    2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST), or total bilirubin levels: > upper limit of normal (ULN).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 703 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, MD, Study Director — Takeda Development Center Asia, Pte Ltd.
Locations (72):
- China (41):
  - Beijing Chao Yang Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The General Hospital of Peoples Armed Police Forces China, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical Univeristy, Beijing, Beijing Municipality
  - Fuzhou General Hospital of Nanjing Military Command, Fuzhou, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat- Sen University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The 2nd Xiangya Hospital Central South University, Changsha, Hu'nan
  - Chenzhou No.1 People's Hospital, Chenzhou, Hu'nan
  - Xiangtan Central Hospital, Xiangtan, Hu'nan
  - Union Hospital of Tongji Medical College of Huazhong Science and Techology University, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Techology, Wuhan, Hubei
  - Peoples Hospital of Wuhan University, Wuhan, Hubei
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Province People's Hospital, Nanjing, Jiangsu
  - Yangzhou 1st Hospital, Yangzhou, Jiangsu
  - No.2 Hospital Affiliated to Jilin University, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University, Jilin, Jilin
  - Jilin central Hospital, Jilin, Jilin
  - Jilin Siping Central Hospital, Siping, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia Hui
  - Ruijin Hospital, Shanghai Jiaotong Uni. School of Med., Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - TongJi Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Sixth Peoples Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The 2nd Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The First Affiated Hospital of Kunming Medical College, Kunming, Yun'nan
  - 2nd Affiliated Hospital, Zhejiang Univ. School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - PLA.The Military General Hospital of Beijing, Beijing
  - Beijing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - 1st Affiliated Hospital of Zhejiang University, Hangzhou
  - The First Affiliated Hospital of NanChang University, Nanchang
  - The Affiliated DrumTower Hospital of Nanjing University, Nanjing
  - Tianjing
- Malaysia (8):
  - Hospital Sultana Bahiyah, Alor Star, Kedah
  - Hospital Universiti Sains Malaysia, Kelantan, Kelantan
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Hospital Queen Elizabeth, Kota Kinabalu, Sabah
  - Hospital Ampang, Ampang, Selangor
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
- South Korea (12):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Gyeonggi-do
  - Kyungpook National University Medical Center, Daegu, Gyeongsangbuk-do
  - Wonkwang University School Of Medicine & Hospital, Iksan-si, Jeollabuk-do
  - Pusan National University Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Marys Hospital, Seoul
- Taiwan (11):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Xiao Y, Qian J, Zhang S, Dai N, Chun HJ, Chiu C, Chong CF, Funao N, Sakurai Y, Eisner JD, Xie L, Chen M. Vonoprazan 10 mg or 20 mg vs. lansoprazole 15 mg as maintenance therapy in Asian patients with healed erosive esophagitis: A randomized controlled trial. Chin Med J (Engl). 2024 Apr 20;137(8):962-971. doi: 10.1097/CM9.0000000000003068. Epub 2024 Mar 29. PMID 38654422

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 64 investigative sites in China, Malaysia, South Korea, and Taiwan from 01 April 2015 to 31 December 2018.
Pre-assignment Details: Participants with a diagnosis of erosive esophagitis were enrolled to receive lansoprazole 30 mg for 4 or 8 weeks (Healing Phase); or vonoprazan 10 mg, 20 mg; or lansoprazole 15 mg once daily for up to 24 weeks (Maintenance Phase).
Period: Overall Study
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg | Lansoprazole 15 mg
Started | 235 | 226 | 242
Completed | 181 | 166 | 180
Not Completed | 54 | 60 | 62
Not completed — Pretreatment Event/Adverse Event | 13 | 11 | 12
Not completed — Major Protocol Deviation | 18 | 25 | 22
Not completed — Lost to Follow-up | 5 | 1 | 4
Not completed — Voluntary Withdrawal | 10 | 18 | 17
Not completed — Lack of Efficacy | 3 | 0 | 3
Not completed — Reason Not Specified | 5 | 5 | 4

BASELINE CHARACTERISTICS:
Population: Randomized set included all randomized participants. The number analyzed is the number of participants with data available for analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg | Lansoprazole 15 mg | Total
Number analyzed (Participants) | 235 | 226 | 242 | 703
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (11.79) | 52.8 (13.02) | 54.0 (12.80) | 52.8 (12.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 61 | 64 | 184
  Male | 176 | 165 | 178 | 519
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 235 | 225 | 242 | 702
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 163 | 159 | 169 | 491
  Malaysia | 24 | 24 | 24 | 72
  Korea, Republic Of | 26 | 23 | 27 | 76
  Taiwan, Province Of China | 22 | 20 | 22 | 64
Height [Mean (Standard Deviation); unit: centimeter (cm)] — Population: The number analyzed is the number of participants with data available for analysis.
  centimeter (cm)
    number analyzed (Participants) | 235 | 225 | 241 | 701
    (all) | 166.7 (8.35) | 166.1 (8.31) | 167.1 (8.01) | 166.7 (8.22)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  kilogram (kg)
    number analyzed (Participants) | 235 | 226 | 240 | 701
    (all) | 70.03 (12.137) | 68.10 (11.314) | 69.19 (11.075) | 69.12 (11.528)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index=weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  kg/m^2
    number analyzed (Participants) | 235 | 225 | 239 | 699
    (all) | 25.10 (3.449) | 24.58 (3.052) | 24.77 (3.475) | 24.82 (3.338)
Smoking Classification [Count of Participants; unit: Participants]
  The Participant Has Never Smoked | 157 | 135 | 147 | 439
  The Participant Is a Current Smoker | 50 | 47 | 55 | 152
  The Participant Is an Ex-smoker | 28 | 44 | 40 | 112
Consumption of Alcohol [Count of Participants; unit: Participants]
  Drink Everyday | 11 | 12 | 16 | 39
  Drink a Couple of Days Per Week | 28 | 19 | 29 | 76
  Drink a Couple of Days Per Month | 53 | 48 | 41 | 142
  Never Drink | 143 | 147 | 156 | 446
Consumption of Caffeine [Count of Participants; unit: Participants]
  Yes | 37 | 34 | 43 | 114
  No | 198 | 192 | 199 | 589
History of H.pylori Eradication Therapy [Count of Participants; unit: Participants]
  Yes (End of Treatment: Within Past 1 Year) | 6 | 9 | 11 | 26
  Yes (End of Treatment: More than 1 Year) | 20 | 19 | 16 | 55
  No | 209 | 198 | 215 | 622
LA Classification (Time of Diagnosis) [Count of Participants; unit: Participants] — Grade A: >/=1 mucosal breaks </=5 mm, none of which extends between the tops of the mucosal folds; Grade B: >/=1 mucosal breaks >5 mm, none of which extends between the tops of two mucosal folds; Grade C: mucosal breaks that extend between the tops of two or more mucosal folds, but which involve <75% of esophageal circumference; Grade D: mucosal breaks which involve >/=75% of esophageal circumference.
  Participants
    Grade A | 91 | 96 | 93 | 280
    Grade B | 94 | 84 | 100 | 278
    Grade C | 42 | 39 | 38 | 119
    Grade D | 8 | 7 | 11 | 26
    Grade A/B | 185 | 180 | 193 | 558
    Grade C/D | 50 | 46 | 49 | 145
Barrett's Mucosa (Baseline) [Count of Participants; unit: Participants]
  Present (3 cm or Greater) | 3 | 0 | 3 | 6
  Present (Less than 3 cm) | 16 | 24 | 16 | 56
  Absent | 212 | 197 | 218 | 627
  Unknown | 4 | 5 | 4 | 13
Esophageal Hiatal Hernia (Baseline) [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    Present (2 cm or Greater): number analyzed (Participants) | 235 | 226 | 241 | 702
    Present (2 cm or Greater) | 27 | 22 | 23 | 72
    Present (Less than 2 cm): number analyzed (Participants) | 235 | 226 | 241 | 702
    Present (Less than 2 cm) | 30 | 22 | 29 | 81
    Absent: number analyzed (Participants) | 235 | 226 | 241 | 702
    Absent | 174 | 179 | 184 | 537
    Unknown: number analyzed (Participants) | 235 | 226 | 241 | 702
    Unknown | 4 | 3 | 5 | 12
HRQoL (EQ-5D-5L) [Mean (Standard Deviation); unit: score on scale] — The Health Related Quality of Life using the EuroQol HRQoL (EQ-5D-5L) has two components: a five-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and a visual analogue scale (VAS) that measures overall health state. Overall scores range from 0 to 1, with lower scores indicating a higher level of dysfunction Population: The number analyzed is the number of participants with data available for analysis.
  score on scale
    number analyzed (Participants) | 226 | 221 | 235 | 682
    (all) | 0.9723 (0.04610) | 0.9723 (0.05252) | 0.9696 (0.06227) | 0.9713 (0.05410)
EQ VAS Score (Baseline) [Mean (Standard Deviation); unit: score on scale] — The EQ visual analogue scale (VAS) records the participant's self-rated health on a 20-cm visual analogue scale ranging from 0 (worst) to 100 (best). Population: The number analyzed is the number of participants with data available for analysis.
  score on scale
    number analyzed (Participants) | 226 | 221 | 235 | 682
    (all) | 88.2 (11.10) | 89.3 (8.85) | 89.4 (9.03) | 89.0 (9.71)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Recurrence of Erosive Esophagitis as Confirmed on Endoscopy After the 24-week Maintenance Phase
Description: Erosive esophagitis recurrence is defined as participants endoscopically confirmed to have erosive esophagitis (Los Angeles [LA] classification grades A to D) during the Maintenance Phase (24 weeks). Grade A: >/=1 mucosal breaks </=5 mm, none of which extends between the tops of the mucosal folds; Grade B: >/=1 mucosal breaks >5 mm, none of which extends between the tops of two mucosal folds; Grade C: mucosal breaks that extend between the tops of two or more mucosal folds, but which involve <75% of esophageal circumference; Grade D: mucosal breaks which involve >/=75% of esophageal circumference.
Time Frame: 24 weeks
Population: Full analysis set included all randomized participants who received at least 1 dose of the Maintenance Phase drug and had at least 1 post-baseline endoscopy, and was based on randomized treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg | Lansoprazole 15 mg
Number analyzed (Participants) | 235 | 226 | 242
percentage of participants | 13.3 [8.684 to 19.084] | 12.3 [7.765 to 18.158] | 25.5 [19.412 to 32.481]

2. Secondary Outcome: Percentage of Participants With Recurrence of Erosive Esophagitis After 12 Weeks of Treatment in the Maintenance Phase
Description: Erosive esophagitis recurrence is defined as endoscopically confirmed to have erosive esophagitis (LA classification grades A to D) during the Maintenance Phase (12 weeks). Grade A: >/=1 mucosal breaks </=5 mm, none of which extends between the tops of the mucosal folds; Grade B: >/=1 mucosal breaks >5 mm, none of which extends between the tops of two mucosal folds; Grade C: mucosal breaks that extend between the tops of two or more mucosal folds, but which involve <75% of esophageal circumference; Grade D: mucosal breaks which involve >/=75% of esophageal circumference.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg | Lansoprazole 15 mg
Number analyzed (Participants) | 235 | 226 | 242
percentage of participants | 27.8 [9.695 to 53.480] | 10.0 [1.235 to 31.698] | 35.0 [15.391 to 59.219]

3. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug whether or not it is considered related to the drug.
Time Frame: From Day 1 to 14 days after the last dose of study medication (up to 26 weeks)
Population: Safety analysis set included all participants who took at least 1 dose of the Maintenance Phase drug and was based on the treatment received in the Maintenance Phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg | Lansoprazole 15 mg
Number analyzed (Participants) | 235 | 226 | 242
Participants | 157 | 156 | 158

4. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Findings
Description: Clinical laboratory safety tests included chemistry, hematology and urinalysis. Number of participants with any markedly abnormal values in laboratory tests collected throughout study is reported. ALT = alanine aminotransferase, AST = aspartate aminotransferase, GGT = gamma-glutamyl transferase, CPK = creatine phosphokinase, BUN = blood urea nitrogen, LLN = lower limit of normal or lower reference limit, ULN = upper limit of normal or upper reference limit, g/L = grams per liter, U/L = units per liter, mmol/L = millimoles per liter, pmol/L = picomoles per liter.
Time Frame: From Day 1 to 14 days after the last dose of study medication (up to 26 weeks)
Population: Safety analysis set included all participants who took at least 1 dose of the Maintenance Phase drug and was based on the treatment received in the Maintenance Phase. The number analyzed is the number of participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg | Lansoprazole 15 mg
Number analyzed (Participants) | 235 | 226 | 242
Participants
  Hematology: Red Blood Cells (>1.2xULN): number analyzed (Participants) | 230 | 219 | 236
  Hematology: Red Blood Cells (>1.2xULN) | 1 | 0 | 1
  Hematology: White Blood Cells (>1.5xULN): number analyzed (Participants) | 230 | 219 | 236
  Hematology: White Blood Cells (>1.5xULN) | 0 | 0 | 1
  Hematology: Hemoglobin (<0.8xLLN): number analyzed (Participants) | 230 | 219 | 236
  Hematology: Hemoglobin (<0.8xLLN) | 1 | 1 | 1
  Hematology: Hematocrit (<0.8xLLN): number analyzed (Participants) | 230 | 219 | 236
  Hematology: Hematocrit (<0.8xLLN) | 0 | 1 | 1
  Hematology: Platelets (<75x10^9/L): number analyzed (Participants) | 230 | 219 | 236
  Hematology: Platelets (<75x10^9/L) | 0 | 1 | 0
  Hematology: Neutrophils (<0.5xLLN): number analyzed (Participants) | 230 | 218 | 235
  Hematology: Neutrophils (<0.5xLLN) | 1 | 0 | 0
  Hematology: Eosinophils (>2xULN): number analyzed (Participants) | 230 | 218 | 235
  Hematology: Eosinophils (>2xULN) | 2 | 2 | 0
  Hematology: Lymphocytes (>1.5xULN): number analyzed (Participants) | 230 | 218 | 235
  Hematology: Lymphocytes (>1.5xULN) | 1 | 0 | 0
  Serum Chemistry: ALT (>3xULN): number analyzed (Participants) | 234 | 222 | 239
  Serum Chemistry: ALT (>3xULN) | 1 | 1 | 0
  Serum Chemistry: AST (>3xULN): number analyzed (Participants) | 234 | 222 | 239
  Serum Chemistry: AST (>3xULN) | 2 | 0 | 2
  Serum Chemistry: GGT (>3xULN): number analyzed (Participants) | 230 | 220 | 236
  Serum Chemistry: GGT (>3xULN) | 4 | 2 | 7
  Serum Chemistry: CK (CPK) (>5xULN): number analyzed (Participants) | 230 | 220 | 236
  Serum Chemistry: CK (CPK) (>5xULN) | 4 | 2 | 3
  Serum Chemistry: Albumin (<25 g/L): number analyzed (Participants) | 230 | 220 | 236
  Serum Chemistry: Albumin (<25 g/L) | 0 | 0 | 1
  Serum Chemistry: Creatinine (>177 umol/L): number analyzed (Participants) | 230 | 220 | 236
  Serum Chemistry: Creatinine (>177 umol/L) | 0 | 0 | 1
  Serum Chemistry: BUN (>10.7 mmol/L): number analyzed (Participants) | 230 | 220 | 236
  Serum Chemistry: BUN (>10.7 mmol/L) | 2 | 4 | 2
  Serum Chemistry: Uric Acid (>0.773 mmol/L): number analyzed (Participants) | 230 | 220 | 236
  Serum Chemistry: Uric Acid (>0.773 mmol/L) | 0 | 1 | 0
  Serum Chemistry: Total Cholesterol (>7.72 mmol/L): number analyzed (Participants) | 230 | 220 | 236
  Serum Chemistry: Total Cholesterol (>7.72 mmol/L) | 2 | 5 | 3
  Serum Chemistry: Triglycerides (>2.5xULN): number analyzed (Participants) | 230 | 220 | 236
  Serum Chemistry: Triglycerides (>2.5xULN) | 2 | 5 | 6
  Serum Chemistry: Glucose (<2.8 mmol/L): number analyzed (Participants) | 230 | 220 | 236
  Serum Chemistry: Glucose (<2.8 mmol/L) | 1 | 0 | 1
  Serum Chemistry: Glucose (>19.4 mmol/L): number analyzed (Participants) | 230 | 220 | 236
  Serum Chemistry: Glucose (>19.4 mmol/L) | 1 | 0 | 0
  Serum Chemistry: Potassium (<3.0 mmol/L): number analyzed (Participants) | 230 | 220 | 236
  Serum Chemistry: Potassium (<3.0 mmol/L) | 0 | 0 | 1
  Serum Chemistry: Sodium (>150 mmol/L): number analyzed (Participants) | 230 | 220 | 236
  Serum Chemistry: Sodium (>150 mmol/L) | 1 | 0 | 0
  Serum Chemistry: Vitamin B12 (<92 pmol/L): number analyzed (Participants) | 230 | 220 | 236
  Serum Chemistry: Vitamin B12 (<92 pmol/L) | 1 | 0 | 3

5. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Number of participants with any markedly abnormal 12-lead ECG findings is reported. bpm = beats per minute, msec = milliseconds, CHG= change from baseline.
Time Frame: From Day 1 to 14 days after the last dose of study medication (up to 26 weeks)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg | Lansoprazole 15 mg
Number analyzed (Participants) | 235 | 226 | 242
Participants
  Heart Rate (<50 bpm): number analyzed (Participants) | 222 | 215 | 227
  Heart Rate (<50 bpm) | 8 | 7 | 4
  Heart Rate (>120 bpm): number analyzed (Participants) | 222 | 215 | 227
  Heart Rate (>120 bpm) | 0 | 1 | 0
  QT Interval (>=460 msec): number analyzed (Participants) | 222 | 215 | 227
  QT Interval (>=460 msec) | 9 | 5 | 8
  QTcF Interval (>= 500, or >= 450 with CHG >= 30): number analyzed (Participants) | 222 | 215 | 227
  QTcF Interval (>= 500, or >= 450 with CHG >= 30) | 8 | 3 | 6

6. Secondary Outcome: Number of Participants With Abnormal Vital Sign Measurements
Description: The percentage of participants with any markedly abnormal vital sign measurements including (body temperature, blood pressure and pulse), mmHg = millimeters of mercury.
Time Frame: From Day 1 to 14 days after the last dose of study medication (up to 26 weeks)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg | Lansoprazole 15 mg
Number analyzed (Participants) | 235 | 226 | 242
Participants
  Body Temperature (<35.6 °Celsius): number analyzed (Participants) | 230 | 221 | 236
  Body Temperature (<35.6 °Celsius) | 6 | 3 | 12
  Body Temperature (>37.7 °Celsius): number analyzed (Participants) | 230 | 221 | 236
  Body Temperature (>37.7 °Celsius) | 0 | 1 | 0
  Systolic Blood Pressure (<85 mmHg): number analyzed (Participants) | 230 | 221 | 236
  Systolic Blood Pressure (<85 mmHg) | 2 | 0 | 0
  Diastolic Blood Pressure (<50 mmHg): number analyzed (Participants) | 230 | 221 | 236
  Diastolic Blood Pressure (<50 mmHg) | 0 | 2 | 1
  Diastolic Blood Pressure (>110 mmHg): number analyzed (Participants) | 230 | 221 | 236
  Diastolic Blood Pressure (>110 mmHg) | 1 | 0 | 0
  Pulse (<50 bpm): number analyzed (Participants) | 230 | 221 | 236
  Pulse (<50 bpm) | 1 | 4 | 3
  Pulse (>120 bpm): number analyzed (Participants) | 230 | 221 | 236
  Pulse (>120 bpm) | 1 | 1 | 0

7. Secondary Outcome: Change From Baseline in Serum Gastrin
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg | Lansoprazole 15 mg
Number analyzed (Participants) | 235 | 226 | 242
pmol/L
  Baseline: number analyzed (Participants) | 230 | 224 | 236
  Baseline | 20.42 (33.969) | 17.97 (21.458) | 21.94 (27.905)
  Change at Week 4: number analyzed (Participants) | 223 | 216 | 231
  Change at Week 4 | 10.09 (37.747) | 22.76 (36.053) | -11.21 (24.651)
  Change at Week 12: number analyzed (Participants) | 207 | 196 | 211
  Change at Week 12 | 14.45 (29.439) | 31.92 (45.127) | -8.76 (24.578)
  Change at Week 24: number analyzed (Participants) | 182 | 172 | 183
  Change at Week 24 | 17.47 (39.847) | 37.60 (47.172) | -7.41 (22.210)

8. Secondary Outcome: Change From Baseline in Serum Pepsinogen I
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg | Lansoprazole 15 mg
Number analyzed (Participants) | 235 | 226 | 242
ug/L
  Baseline: number analyzed (Participants) | 232 | 225 | 237
  Baseline | 287.1 (249.41) | 276.3 (203.46) | 303.3 (253.76)
  Change at Week 4: number analyzed (Participants) | 227 | 218 | 232
  Change at Week 4 | 40.5 (266.92) | 139.8 (269.08) | -112.3 (245.22)
  Change at Week 12: number analyzed (Participants) | 210 | 199 | 211
  Change at Week 12 | -3.1 (267.65) | 89.9 (285.05) | -123.5 (252.45)
  Change at Week 24: number analyzed (Participants) | 182 | 173 | 183
  Change at Week 24 | 5.9 (289.91) | 55.4 (279.65) | -103.9 (218.80)

9. Secondary Outcome: Change From Baseline in Serum Pepsinogen II
Time Frame: Baseline and Weeks 4, 12 and 24
Population: Safety analysis set included all participants who took at least 1 dose of the Maintenance Phase drug and was based on the treatment received in the Maintenance Phase.The number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg | Lansoprazole 15 mg
Number analyzed (Participants) | 235 | 226 | 242
ug/L
  Baseline: number analyzed (Participants) | 233 | 224 | 237
  Baseline | 22.9 (22.42) | 22.1 (17.40) | 24.6 (23.83)
  Change at Week 4: number analyzed (Participants) | 228 | 219 | 231
  Change at Week 4 | 3.8 (27.34) | 16.5 (25.56) | -10.9 (23.98)
  Change at Week 12: number analyzed (Participants) | 211 | 199 | 211
  Change at Week 12 | -1.6 (24.02) | 9.0 (26.40) | -10.9 (24.41)
  Change at Week 24: number analyzed (Participants) | 184 | 173 | 183
  Change at Week 24 | -0.6 (27.23) | 5.8 (25.59) | -8.7 (19.61)

ADVERSE EVENTS:
Time Frame: Up to 26 weeks
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Vonoprazan 10 mg | Vonoprazan 20 mg | Lansoprazole 15 mg
All-Cause Mortality (participants affected / at risk) | 0/235 | 0/226 | 1/242
Serious Adverse Events (participants affected / at risk) | 10/235 | 8/226 | 12/242
Other Adverse Events (participants affected / at risk) | 81/235 | 79/226 | 79/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan 10 mg (N=235) | Vonoprazan 20 mg (N=226) | Lansoprazole 15 mg (N=242)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 0
Iridocyclitis (Eye disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Typhoid fever (Infections and infestations) | 0 | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 2 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Laryngeal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vonoprazan 10 mg (N=235) | Vonoprazan 20 mg (N=226) | Lansoprazole 15 mg (N=242)
Diarrhoea (Gastrointestinal disorders) | 15 | 21 | 17
Dyspepsia (Gastrointestinal disorders) | 18 | 10 | 12
Gastric polyps (Gastrointestinal disorders) | 11 | 12 | 8
Abdominal distension (Gastrointestinal disorders) | 5 | 6 | 13
Upper respiratory tract infection (Infections and infestations) | 30 | 29 | 21
Nasopharyngitis (Infections and infestations) | 12 | 12 | 11
Alanine aminotransferase increased (Investigations) | 13 | 9 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT02388737/SAP_000.pdf
  • Study Protocol (2016-11-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT02388737/Prot_001.pdf